CLINICAL TRIAL: NCT06825715
Title: Multilevel Veteran-centric Intervention to Improve Precision Oncology
Brief Title: Multilevel Intervention for Precision Oncology
Acronym: MIPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Madison Health Care (Unknown); VA Pittsburgh Healthcare System (U.S. Federal Agency); Martinsburg VA Medical Center (Unknown); VA Eastern Oklahoma Health Care (Unknown); New Orleans VA Medical Center (Unknown); Northport VA Medical Center (Unknown); Fargo VA Medical Center (U.S. Federal Agency); VA Iron Mountain Health Care (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 22-169
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Advanced Cancers of the Prostate; Cancers of the Lung

STUDY DESIGN:
Intervention Model Description: Multilevel intervention with components of patient education, provider audit/feedback, and change in electronic medical record test order and results return.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- During intervention period (Experimental): All sites will receive the 3 level intervention of patient education, provider audit/feedback, and EMR order change.
  Interventions: Other: Multilevel intervention

INTERVENTIONS:
Other: Multilevel intervention — 3 components: patient education video, provider audit/feedback, and EMR ordering change

SUMMARY:
The investigators are rolling out a 3 level intervention designed to improve the use of Precision Oncology at 8 VA medical centers. The 3 components of the intervention are 1: a short educational video for patients, 2: audit and feedback to providers on their Precision Oncology practice patterns, and 3: a change in the electronic medical record to make it easier to order and review results of Precision Oncology tests.

DETAILED DESCRIPTION:
Background: Precision oncology (PO), the use of molecular testing to identify tumor specific abnormalities which facilitate targeted therapy, is proven to extend lives and improve quality of life for patients with cancer. Extensive study, however, documents that up to 50% of patients in the VA, especially those with adverse social determinants of health (older age, rural), do not receive guideline recommended PO.

Methodology: Building on the investigators' previous analyses, and the Theoretical Domains Framework, the investigators designed a mixed-methods type I hybrid effectiveness-implementation study of a multilevel intervention (MLI) to improve the use of PO. The MLI will be instituted for veterans with advanced cancers of the colon, lung, and prostate, as well as providers at 8 sites, chosen to represent diversity at the level of rurality, geographic region, cancer volume, and mode of delivery (virtual/in-person). The patient intervention is a 5-minute educational module accessible by QR code. The provider intervention is a 45-minute academic detailing session, as well as individualized audit and feedback on practice patterns. The facility level intervention is a previously piloted integration of PO ordering, interdepartmental communication, and results return into the primary electronic medical record via a consult function. The primary efficacy outcome is the rate of molecular testing/eligible veterans. Validated survey measures will be used for stakeholder engagement. The process evaluation employs a mixed methods approach based in the RE-AIM framework, which includes quantitative analyses of collected data, and interviews of patients and providers. The statistical design is a randomized stepped-wedge trial over 3 years which retains control data from across all sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the VA with cancer of the lung or prostate who are seen in the oncology clinic

Exclusion Criteria:

* Cancer that did not originate in the prostate or the lung

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2653 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Use of molecular testing | 3 years
  Proportion of eligible patients with lung and prostate cancer who have next generation sequencing molecular testing

SECONDARY OUTCOMES:
Use of targeted therapy | 3 years
  Proportion of patients with actionable molecular alterations who have targeted therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Becker, MD, Principal Investigator — VA NY Harbor Healthcare System, New York, NY
Locations (1):
- VA NY Harbor Healthcare System, New York, NY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No